CLINICAL TRIAL: NCT02141295
Title: A Phase II, Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of RO5520985 (Vanucizumab) Plus FOLFOX Versus Bevacizumab Plus FOLFOX in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: A Study Comparing the Efficacy and Safety of Vanucizumab and FOLFOX With Bevacizumab and FOLFOX in Participants With Untreated Metastatic Colorectal Cancer
Acronym: McCAVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP29262; 2013-005108-32 (EudraCT Number)
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Leucovorin; Oxaliplatin; vanucizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 (Induction): Vanucizumab + mFOLFOX-6 (Experimental): Participants will receive vanucizumab at a dose of 2000 milligram (mg) as intravenous (IV) infusion; oxaliplatin at a dose of 85 mg per meter-squared (mg/m^2) as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks for up to 8 cycles (approximately 4 months).
  Interventions: Drug: 5-FU; Drug: Folinic acid; Drug: Oxaliplatin; Drug: Vanucizumab
- Part 1 (Maintenance): Vanucizumab + 5-FU + Folinic acid (Experimental): Participants will receive vanucizumab at a dose confirmed during induction as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks until disease progression, unacceptable toxicities, consent withdrawal or Investigator's decision for a maximum of 24 months.
  Interventions: Drug: 5-FU; Drug: Folinic acid; Drug: Vanucizumab
- Part 2 (Induction): Bevacizumab + mFOLFOX-6 (Active Comparator): Participants will receive bevacizumab at a dose of 5 milligram per kilogram (mg/kg) as IV infusion; oxaliplatin at a dose of 85 mg/m^2 as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks for up to 8 cycles (approximately 4 months).
  Interventions: Drug: 5-FU; Drug: Bevacizumab; Drug: Folinic acid; Drug: Oxaliplatin
- Part 2 (Induction): Vanucizumab + mFOLFOX-6 (Experimental): Participants will receive vanucizumab at a dose confirmed during part 1 as IV infusion; oxaliplatin at a dose of 85 mg/m^2 as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks for up to 8 cycles (approximately 4 months).
  Interventions: Drug: 5-FU; Drug: Folinic acid; Drug: Oxaliplatin; Drug: Vanucizumab
- Part 2 (Maintenance): Bevacizumab + 5-FU + Folinic acid (Active Comparator): Participants will receive bevacizumab at a dose of 5 mg/kg as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks until disease progression, unacceptable toxicities, consent withdrawal or Investigator's decision for a maximum of 24 months.
  Interventions: Drug: 5-FU; Drug: Bevacizumab; Drug: Folinic acid
- Part 2 (Maintenance): Vanucizumab + 5-FU + Folinic acid (Experimental): Participants will receive vanucizumab at a dose confirmed during part 1 as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks until disease progression, unacceptable toxicities, consent withdrawal or Investigator's decision for a maximum of 24 months.
  Interventions: Drug: 5-FU; Drug: Folinic acid; Drug: Vanucizumab

INTERVENTIONS:
Drug: 5-FU — 5-FU will be administered according to dose and schedule described in respective arm.
Drug: Bevacizumab — Bevacizumab will be administered according to dose and schedule described in respective arm.
  Other Names: Avastin
  Arms: Part 2 (Induction): Bevacizumab + mFOLFOX-6; Part 2 (Maintenance): Bevacizumab + 5-FU + Folinic acid
Drug: Folinic acid — Folinic acid will be administered according to dose and schedule described in respective arm.
Drug: Oxaliplatin — Oxaliplatin will be administered according to dose and schedule described in respective arm.
  Arms: Part 1 (Induction): Vanucizumab + mFOLFOX-6; Part 2 (Induction): Bevacizumab + mFOLFOX-6; Part 2 (Induction): Vanucizumab + mFOLFOX-6
Drug: Vanucizumab — Vanucizumab will be administered according to dose and schedule described in respective arm.
  Other Names: RO5520985
  Arms: Part 1 (Induction): Vanucizumab + mFOLFOX-6; Part 1 (Maintenance): Vanucizumab + 5-FU + Folinic acid; Part 2 (Induction): Vanucizumab + mFOLFOX-6; Part 2 (Maintenance): Vanucizumab + 5-FU + Folinic acid

SUMMARY:
This is a Phase 2 multicenter, randomized, parallel arms, double-blind study of vanucizumab to evaluate the efficacy and safety of vanucizumab in combination with oxaliplatin, folinic acid, and 5-fluorouracil (5-FU) (mFOLFOX-6) versus bevacizumab (Avastin) + mFOLFOX-6 in participants with previously untreated metastatic colorectal cancer (mCRC). The study consists of 2 parts: a safety run-in open-label, single-arm part (Part 1) and a randomized, parallel-arms, double-blind part (Part 2). During Part 1 at least 6 eligible participants will receive 2000 milligrams (mg) vanucizumab every 2 weeks + mFOLFOX-6 in order to confirm the dose and schedule that will be used in Part 2. In Part 2, all eligible participants will be randomized in a ratio of 1:1 to receive either mFOLFOX-6 + vanucizumab or mFOLFOX-6 + bevacizumab. Study treatment (induction and maintenance) will be given on Day 1 of each 14-day cycle. Induction therapy will consist of up to 8 cycles of mFOLFOX-6 plus either bevacizumab or vanucizumab. Maintenance therapy will consist of 5-fluorouracil and folinic acid plus either vanucizumab or bevacizumab for up to 24 months or until disease progression, unacceptable toxicity, Investigator decision or consent withdrawal, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed mCRC not amenable to potentially curative resection with at least one measurable metastatic lesion, as defined by RECIST v1.1
* Eastern Cooperative Oncology Group (World Health Organization) performance status of 0 or 1
* Adequate hematologic, liver, coagulation, renal, and cardiovascular function
* Recovery from all reversible AEs of previous medical therapies to baseline or National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade 1, except for alopecia (any grade)
* Negative serum pregnancy test within 7 days prior to starting study treatment in premenopausal women and women less than (< 2) years after the onset of menopause

Exclusion Criteria:

* Any prior systemic therapy (including chemotherapy, antibody therapy, tyrosine kinase inhibitors, immunotherapy, hormonal therapy) before Day 1 of Cycle 1 for treatment of mCRC
* Malignancies other than CRC within 5 years prior to randomization, except for those with a minimal risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ treated surgically with curative intent
* Radiotherapy within 28 days and abdominal/ pelvic radiotherapy within 60 days prior to Day 1 of Cycle 1, except palliative radiotherapy to bone lesions within 7 days prior to Day 1 of Cycle 1
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to Day 1 of Cycle
* Pregnant or lactating women
* Symptomatic central nervous system (CNS) metastases or carcinomatous meningitis. Asymptomatic patients must be clinically stable with regard to their CNS/ meningeal metastatic involvement, have completed previous therapy (including radiation and/ or surgery) at least 4 weeks prior to study drug administration, are not receiving steroid therapy or taper, and are not receiving anti-convulsive medication for any CNS involvement
* Active infection requiring IV antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs (NSAIDs), inhaled corticosteroids, or the equivalent of less than or equal to (</=) 10 mg/day prednisone
* Sensory peripheral neuropathy greater than or equal to (>/=) Grade 2
* Significant cardiovascular or cerebrovascular disease within 6 months prior to Day 1 of Cycle 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation
* Current use of anticoagulants at therapeutic doses within 7 days prior to study drug administration. Prophylactic use of unfractioned heparin or low molecular weight heparin is permitted
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of Cycle 1 or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to Day 1 of Cycle 1
* History of intra-abdominal inflammatory process within 6 months prior to Day 1 of Cycle 1 including but not limited to peptic ulcer disease, diverticulitis, or colitis
* Colonic prosthesis (stent) implant in place
* History of abdominal or tracheo-oesophageal fistula or gastrointestinal (GI) perforation or intra abdominal abscess within 6 months prior to Day 1 of Cycle 1
* History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or a requirement for routine parenteral hydration, parenteral nutrition, or tube feeding within 6 months prior to Day 1 of Cycle 1
* Chronic daily treatment with NSAID (occasional use for the symptomatic relief of medical conditions, for example headache or fever is allowed)
* Chronic daily treatment with corticosteroids (dose > 10 mg/day methylprednisolone equivalent) excluding inhaled steroids
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Metastatic disease that involve major airways or blood vessels, or centrally located mediastinal tumor masses (< 30 millimeter from the carina) of large volume
* History of bronchopulmonary hemorrhage NCI CTCAE >/= Grade 2 within 2 months prior to randomization
* Severe, nonhealing or open wound, active ulcer, or untreated bone fracture
* Known dihydropyrimidine dehydrogenase deficiency or thymidylate synthase gene polymorphism predisposing the patient for 5-FU toxicity
* Any other condition, diseases, metabolic dysfunction, active or uncontrolled infections/inflammation, physical examination finding, mental status or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates participation in the clinical study due to safety concerns, compliance with clinical study procedures or that may affect the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- United States (14):
  - Alabama Oncology, Birmingham, Alabama
  - Arizona Clinical Research Ctr, Tucson, Arizona
  - California Cancer Associates for Research & Excellence, Inc., Encinitas, California
  - Fresno cCare, Fresno, California
  - University of California San Diego Medical Center, La Jolla, California
  - Va Greater Los Angeles Healthcare System, Sepulveda, California
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Ctr for Cancer and Blood Disorders, Fort Worth, Texas
  - Cancer Therapy & Research Center, San Antonio, Texas
  - Northern Utah Associates, Ogden, Utah
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Monash Medical Centre-Moorabbin Campus, Clayton, Victoria
- Austria (2):
  - Salzburger Landeskliniken LKH, Salzburg
  - Oö. Gesundheits- und Spitals-AG/LKH Steyr, Steyr
- Imeldaziekenhuis, Bonheiden, Belgium
- France (2):
  - Centre Paul Papin, Angers
  - Institut De Cancerologie De L'Ouest; Medical Oncology, Saint-Herblain
- Spain (12):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Reina Sofia; Servicio de Oncologia, Córdoba, Cordoba
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - HM Sanchinarro - CIOCC; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (5):
  - Aberdeen Royal Infirmary; Medical Oncology Dept, Aberdeen
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Maidstone Hospital, Maidstone
  - Queen's Hospital; Oncology, Romford
  - The Royal Marsden Hospital, Sutton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with previously untreated metastatic colorectal cancer (mCRC) as defined by RECIST v1.1 were enrolled globally from 7 countries.
Groups:
- Safety Run-In: 8 eligible participants received 2000 milligrams (mg) vanucizumab + mFOLFOX-6 every two weeks for up to 8 cycles in order to confirm the dose and schedule for the randomized part.
- Vanucizumab + mFOLFOX-6: In the induction therapy participants received vanucizumab at a dose of 2000 mg as IV infusion; oxaliplatin at a dose of 85 mg/m^2 as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks for up to 8 cycles (approximately 4 months). Subsequently, in the maintenance therapy participants received vanucizumab at a dose of 2000 mg as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks until disease progression, unacceptable toxicities, consent withdrawal or Investigator's decision for a maximum of 24 months.
- Bevacizumab + mFOLFOX-6: In the induction therapy participants received bevacizumab at a dose of 5 milligram per kilogram (mg/kg) as IV infusion; oxaliplatin at a dose of 85 mg/m^2 as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks for up to 8 cycles (approximately 4 months). Subsequently, in the maintenance therapy participants received bevacizumab at a dose of 5 milligram per kilogram (mg/kg) as IV infusion; folinic acid at a dose of 400 mg/m^2 as IV infusion; and 5-FU at a dose of 400 mg/m^2 as starting IV bolus followed by 2400 mg/m^2 as IV infusion every 2 weeks until disease progression, unacceptable toxicities, consent withdrawal or Investigator's decision for a maximum of 24 months.
Period: Overall Study
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6
Started | 8 | 94 | 95
Completed | 2 | 0 | 0
Not Completed | 6 | 94 | 95
Not completed — Adverse Event | 1 | 18 | 11
Not completed — Physician Decision | 2 | 19 | 14
Not completed — Study terminated by sponsor | 0 | 6 | 6
Not completed — Non-compliance | 0 | 1 | 0
Not completed — Progressive disease | 3 | 32 | 50
Not completed — Reason not specified | 0 | 9 | 10
Not completed — Withdrawal by Subject | 0 | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6 | Total
Number analyzed (Participants) | 8 | 94 | 95 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.8) | 62.7 (11.0) | 62.3 (10.6) | 62.5 (0.2)
Age, Customized [Number; unit: Participants]
  Adults (18-64 years) | 4 | 48 | 53 | 105
  From 65-84 years | 4 | 46 | 42 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 38 | 57 | 98
  Male | 5 | 56 | 38 | 99

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS), Time to Event
Description: Efficacy of vanucizumab was evaluated in terms of PFS as Investigator-Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). PFS was defined as the time between randomization and the date of first documented disease progression or death from any cause on study, whichever occurred first. Death on study was defined as death from any cause within 30 days of the last study treatment.
Time Frame: Baseline, every 8 weeks, up to approximately 29 months
Population: This analysis was based on the ITT population, which consisted of all participants who were randomized (Part II only) and received any amount of the study treatment (5 FU/folinic acid, oxaliplatin, bevacizumab, or vanucizumab) in the bevacizumab + mFOLFOX-6 and vanucizumab + mFOLFOX-6 arms. Participants in the safety-run in were not included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 94 | 95
days | 338.0 [312.0 to 381.0] | 309.0 [284.0 to 352.0]
Statistical Analysis 1: Comparison: Vanucizumab + mFOLFOX-6 vs Bevacizumab + mFOLFOX-6; Kaplan-Meier methods were used to estimate median PFS for each treatment arm and the 95% CIs for median PFS were computed using the Brookmeyer and Crowley method. The stratified Cox proportional hazard was used to estimate the hazard ratio (i.e., the magnitude of the treatment effect) and the corresponding 95% confidence interval. The stratification factors are number of metastatic sites (1 vs. >1) and country/region (USA vs rest of the world); Test type: Other; p = 0.6753, Regression, Cox — log-rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.60 to 1.39]

2. Secondary Outcome: Percentage of Participants With Objective Response (ORR) as Assessed Using RECIST v. 1.1
Description: Efficacy of vanucizumab was evaluated in terms of Percentage of Participants With ORR as Investigator-Assessed Using RECIST v. 1.1. Best Overall Confirmed Response.
Time Frame: Baseline (within 28 days prior to Day 1), then every 8 weeks until progressive disease (PD), start of other anticancer therapy, withdrawal of consent, or death (up to approximately 29 months)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 8 | 94 | 95
Percentage of Participants | 62.5 [34.3 to 90.6] | 43.6 [33.59 to 53.64] | 51.6 [41.53 to 61.63]

3. Secondary Outcome: Duration of Objective Response, as Assessed Using RECIST v. 1.1
Description: Efficacy of vanucizumab was evaluated in terms of duration of objective response as assessed using RECIST v. 1.1. This was computed using the PFS definition with death on study (deaths that occurred outside the 30 days window from the last study treatment are excluded).
Time Frame: Baseline (within 28 days prior to Day 1), then every 8 weeks until PD, start of other anticancer therapy, withdrawal of consent, or death (up to approximately 29 months)
Population: This analysis was based on the ITT population, which consisted of all participants in the bevacizumab + mFOLFOX-6 and vanucizumab + mFOLFOX-6 arms. Participants in the safety-run in were not included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 94 | 95
days | 342 [274 to 510] | 304 [220 to 366]

4. Secondary Outcome: Overall Survival (OS)
Description: Efficacy of vanucizumab was evaluated in terms of OS as the time from randomization until death from any cause. 99999 = data not estimable due to the low number of deaths.
Time Frame: Baseline until death from any cause (maximum up to approximately 3.5 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 94 | 95
days | 746.0 [687.0 to NA] — Value is not estimable due to an insufficient number of participants with the event prior to study termination. | NA [723.0 to NA] — Value is not estimable due to an insufficient number of participants with the event prior to study termination.
Statistical Analysis 1: Comparison: Vanucizumab + mFOLFOX-6 vs Bevacizumab + mFOLFOX-6; Kaplan-Meier methods were used to estimate median OS for each treatment arm and the 95% CIs for median OS were computed using the Brookmeyer and Crowley method. The stratified Cox proportional hazard was used to estimate the hazard ratio (i.e., the magnitude of the treatment effect) and the corresponding 95% confidence interval. The stratification factors are number of metastatic sites (1 vs. >1) and country/region (USA vs rest of the world); Test type: Other; p = 0.5740, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.49 to 1.49]

5. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Safety is evaluated in terms of percentage of participants with at least one serious adverse event and percentage of participants with at least one adverse event.
Time Frame: Up to approximately 29 months
Population: n for the vanucizumab + mFOLFOX-6 arm changed from 94 to 93 due to the withdrawal of a participant that was randomized to this arm, but received only chemotherapy before leaving the study. This participant is included in the ITT population but not in the safety population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6
Number analyzed (Participants) | 8 | 93 | 95
Percentage of Participants
  Serious Adverse events | 37.5 | 49.5 | 43.2
  Adverse events | 100 | 100.0 | 100.0

6. Secondary Outcome: Number of Participants With Human Anti-human Antibodies (HAHAs) Against Vanucizumab
Description: Safety is evaluated in terms of number of participants with Human Anti-human Antibodies (HAHAs) Against Vanucizumab.
Time Frame: End of study (EoS, within 28 to 42 days after last dose, latest at 29 months)
Population: Endpoint includes only arms in which the participants received vanucizumab. n for the vanucizumab + mFOLFOX-6 arm changed from 94 to 93 due to the withdrawal of a participant that was randomized to this arm, but received only chemotherapy before leaving the study. This participant is included in the ITT population but not in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 8 | 93
Participants | 2 | 1

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of AUC
Time Frame: Cycles 1 and 8 of parts 1 and 2
Population: This endpoint was only reported for arms in which the participants received vanucizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ug/ml
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 7 | 77
hr*ug/ml
  Cycle 1 | 73600 (20.7) | 63500 (27.2)
  Cycle 8: number analyzed (Participants) | 3 | 45
  Cycle 8 | 112000 (11.2) | 82100 (31.6)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of Cmax
Time Frame: Cycles 1 and 8 of parts 1 and 2
Population: This endpoint was only reported for arms in which the participants received vanucizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 8 | 93
ug/ml
  Cycle 1 | 463 (18.5) | 500 (26.3)
  Cycle 8: number analyzed (Participants) | 6 | 64
  Cycle 8 | 685 (17.6) | 794 (38.2)

9. Secondary Outcome: Minimum Observed Plasma Concentration (Clast) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of Clast
Time Frame: Cycles 1 and 8 of parts 1 and 2
Population: Data were collected and analyzed for the reported arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 93
ug/ml
  Cycle 1 | 103 (67.2)
  Cycle 8: number analyzed (Participants) | 64
  Cycle 8 | 361 (39.8)

10. Secondary Outcome: Time to Reach Cmax (Tmax) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of Tmax
Time Frame: Cycles 1 and 8 of parts 1 and 2
Population: This endpoint was only reported for arms in which the participants received vanucizumab.
Measure: Median (Full Range); unit: hr
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 8 | 93
hr
  Cycle 1 | 2.79 [1.50 to 7.67] | 2.05 [1.0 to 26.1]
  Cycle 8: number analyzed (Participants) | 6 | 64
  Cycle 8 | 4.04 [0.5 to 5.25] | 1.58 [0.5 to 4.77]

11. Secondary Outcome: Plasma Terminal Half-Life (t1/2) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of t1/2, values are reported for cycle 8 of both part 1 (safety run-in) and part 2 of the study.
Time Frame: Cycle 8
Population: This endpoint was only reported for arms in which the participants received vanucizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 3 | 37
hr | 202 (12.4) | 157 (30.3)

12. Secondary Outcome: Plasma Clearance at Steady State (CLss) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of CLss, values are reported for cycle 8 of both part 1 (safety run-in) and part 2 of the study.
Time Frame: Cycle 8
Population: This endpoint was only reported for arms in which the participants received vanucizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml/hr
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 3 | 37
ml/hr | 15.3 (26.7) | 18.0 (29.0)

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of Vss, values are reported for cycle 8 of both part 1 (safety run-in) and part 2 of the study.
Time Frame: Cycle 8
Population: This endpoint was only reported for arms in which the participants received vanucizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ml
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 3 | 37
ml | 4400 (25.1) | 4140 (29.7)

14. Secondary Outcome: Cmax Accumulation Ratio (AR) of Vanucizumab
Description: PK profile of vanucizumab was evaluated in terms of Cmax Ratio, values are reported for cycle 8 of both part 1 (safety run-in) and part 2 of the study.
Time Frame: Cycle 8
Population: This endpoint was only reported for arms in which the participants received vanucizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6
Number analyzed (Participants) | 5 | 64
Ratio | 1.51 (27.2) | 1.63 (36.2)

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose of study drug (maximum treatment time = approximately 29 months).
Description: n for the vanucizumab + mFOLFOX-6 arm changed from 94 to 93 due to the withdrawal of a participant that was randomized to this arm, but received only chemotherapy before leaving the study. This participant is included in the ITT population but not in the safety population.
Arm/Group | Safety Run-In | Vanucizumab + mFOLFOX-6 | Bevacizumab + mFOLFOX-6
All-Cause Mortality (participants affected / at risk) | 3/8 | 24/93 | 27/95
Serious Adverse Events (participants affected / at risk) | 3/8 | 46/93 | 41/95
Other Adverse Events (participants affected / at risk) | 8/8 | 91/93 | 94/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In (N=8) | Vanucizumab + mFOLFOX-6 (N=93) | Bevacizumab + mFOLFOX-6 (N=95)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 4 (8)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumor obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Vasospasm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In (N=8) | Vanucizumab + mFOLFOX-6 (N=93) | Bevacizumab + mFOLFOX-6 (N=95)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (7) | 12 (19)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (6) | 40 (52) | 43 (63)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 4 (6) | 8 (9)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 4 (5) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 27 (33) | 22 (22)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 7 (8) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 6 (9) | 14 (15)
Constipation (Gastrointestinal disorders) | 3 (5) | 26 (36) | 31 (52)
Diarrhoea (Gastrointestinal disorders) | 6 (8) | 56 (107) | 57 (133)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 11 (15) | 8 (12)
Flatulence (Gastrointestinal disorders) | 0 (0) | 5 (6) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 52 (93) | 55 (98)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 15 (25) | 11 (15)
Vomiting (Gastrointestinal disorders) | 1 (1) | 31 (40) | 29 (46)
Asthenia (General disorders) | 3 (6) | 41 (89) | 42 (129)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 5 (5) | 3 (3)
Fatigue (General disorders) | 1 (1) | 26 (33) | 23 (28)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 4 (6) | 23 (42) | 31 (68)
Oedema peripheral (General disorders) | 3 (5) | 11 (15) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 17 (24) | 18 (22)
Temperature intolerance (General disorders) | 1 (1) | 11 (15) | 10 (16)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 8 (9) | 9 (12)
Oral candidiasis (Infections and infestations) | 1 (1) | 5 (5) | 1 (2)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 14 (15)
Urinary tract infection (Infections and infestations) | 2 (3) | 11 (12) | 10 (14)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 19 (26) | 13 (18)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (7) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 9 (9)
Platelet count decreased (Investigations) | 0 (0) | 10 (25) | 4 (6)
Weight decreased (Investigations) | 0 (0) | 12 (13) | 13 (13)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 29 (45) | 33 (67)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 9 (13) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (10)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 9 (10) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4) | 8 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (9) | 16 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 5 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (12) | 7 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (11) | 8 (12)
Pain in extremitiy (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 6 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 2 (4)
Aphonia (Nervous system disorders) | 0 (0) | 5 (5) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 11 (16) | 12 (17)
Dysaesthesia (Nervous system disorders) | 1 (3) | 15 (32) | 22 (79)
Dysgeusia (Nervous system disorders) | 5 (6) | 16 (16) | 22 (26)
Headache (Nervous system disorders) | 2 (2) | 15 (16) | 19 (30)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (8) | 18 (31) | 28 (66)
Neurotoxicity (Nervous system disorders) | 0 (0) | 8 (14) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 15 (17) | 17 (24)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4) | 33 (83) | 28 (72)
Anxiety (Psychiatric disorders) | 1 (1) | 9 (9) | 8 (8)
Depression (Psychiatric disorders) | 1 (1) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 11 (11) | 12 (13)
Dysuria (Renal and urinary disorders) | 0 (0) | 5 (5) | 6 (8)
Proteinuria (Renal and urinary disorders) | 1 (5) | 12 (15) | 10 (17)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (12) | 10 (13)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 13 (13) | 9 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (12) | 10 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 20 (27) | 28 (36)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 7 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 14 (14)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (14) | 16 (23)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (8) | 8 (10)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (7) | 4 (5)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (9) | 42 (75) | 27 (50)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT02141295/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT02141295/SAP_001.pdf